CLINICAL TRIAL: NCT05595577
Title: Improving Exercise Capacity With a Tailored Physical Activity Intervention in Lymphoma and Breast Cancer Patients Undergoing Treatment
Brief Title: Improving Exercise Capacity With a Tailored Physical Activity Intervention
Acronym: PALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00087763; 4R33CA226960-03 (NIH); WFBCCC 98622 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Non Hodgkin Lymphoma; Heart; Functional Disturbance; Hodgkin Lymphoma; Quality of Life; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Exercise capability; Brain activity
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Breast Neoplasms | interventions — Exercise; Exercise Test; Magnetic Resonance Imaging; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All images will be processed offline by an image analyst blinded to study group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Physical Activity Intervention (Experimental): Participants will have the ability to attend one to two training sessions per week and 1-2 sessions per week at home (the 4th level of our multi-level intervention) or the location site using the Trainerize application to deliver the exercise prescription.
  Interventions: Other: Exercise with Trainerize application; Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: MRI scan; Behavioral: Quality of Life Questionnaires; Behavioral: Cognitive and Brain Function Questionnaires; Other: Blood draws
- Healthy Living Intervention (Control Arm) (Experimental): Participants randomized to the control arm will participate in organized health workshops. Each session will last 60 minutes and will be offered on location and virtually (e.g., Zoom) over 6 months. Participants will meet once a week for the first 4 weeks, biweekly for 3 months, and once a month for the last 2 months for a total of 12 sessions.
  Interventions: Diagnostic Test: Cardiopulmonary exercise testing; Diagnostic Test: MRI scan; Behavioral: Quality of Life Questionnaires; Behavioral: Cognitive and Brain Function Questionnaires; Other: Blood draws

INTERVENTIONS:
Other: Exercise with Trainerize application — 1-2 sessions per week consisting of slow 15 minute aerobic warm, 20 minutes of strength training, 15 minutes progressive intensity aerobic exercise and 10 minute cool down (stretching/toning) with elastic bands.
  Arms: Physical Activity Intervention
Diagnostic Test: Cardiopulmonary exercise testing — Maximal peak VO2 (to monitor the body's oxygen consumption) and 6-minute exercise walking test.
Diagnostic Test: MRI scan — Images of the heart will be taken.
Behavioral: Quality of Life Questionnaires — Participants will be asked to complete several questionnaires that will measure fatigue, general health, social determinants of health, cognitive function (tasks that assess memory, ability to count, etc.) and physical activity. The questionnaires will take 15-40 minutes to complete.
Behavioral: Cognitive and Brain Function Questionnaires — Participants will be asked to complete several questionnaires that will measure fatigue, general health, social determinants of health, cognitive function (tasks that assess memory, ability to count, etc.) and physical activity. The questionnaires will take 15-40 minutes to complete.
Other: Blood draws — Approximately 2 teaspoons of blood withdrawn from either a vein in your arm or a currently placed central line port-a-cath. A portion of blood from each visit will be used to collect information about blood cell count.

SUMMARY:
The purpose of this research is to test whether participating in either a physical activity intervention or a series of educational classes will help to preserve exercise capability, heart function, brain-based activities (like memory), and quality of life.

Participants will be randomized to 1 of 2 pathways:

* First pathway consists of organized health workshops. These workshops are intended to provide information on topics such as proper nutrition, management of stress, sleep practices, and emphasis on a healthy lifestyle that may help the participants through cancer treatment. This pathway will also test whether stretching may help participants through cancer treatment.
* Second pathway participants will take part in some unsupervised and some potentially supervised moderate activity sessions each week throughout participants' cancer treatment to take place either remotely or in person, depending on availability of facilities at the time visits are scheduled.

DETAILED DESCRIPTION:
Primary Objective: To determine if a >10% difference exists in the % change (i.e., 2.06 ml/kg/min difference) in peak VO2 (volume or amount of oxygen your body consume) from baseline to 6 months of intervention between participants receiving the Physical Activity Intervention (PAI) versus Healthy Living Intervention (HLI).

Secondary Objectives:

* To determine if a >10% difference exists in the % change in peak exercise cardiac output, calculated A-VO2 difference, and pre-exercise measures of left ventricular function from baseline to 6 months of intervention between participants receiving the PAI versus HLI.
* Among these same participants, 1) to compare PAI and HLI groups on their baseline to 3 & 6 months after initiating cancer treatment changes in 6-minWD, Health-Related Quality of Life (HRQOL), fatigue, strength, physical activity, cognitive & physical function, 2) to determine the relationships between the 6-month time-dependent changes in these and peak VO2; and 3) to examine whether time-dependent changes in peak exercise cardiac output and/or calculated arteriovenous oxygen difference are associated with similar time-dependent changes in peak VO2.
* Assess physical activity engagement via accelerometry.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible, participants must meet all of the following criteria:

* Individuals aged 18- 85 years
* Diagnosed with stage I-IV Hodgkin's or non-Hodgkin's lymphoma or stage I-III breast cancer
* Expected to receive an anthracycline based chemotherapeutic regimen or other potentially cardiotoxic cancer therapies (e.g. chemotherapy regimens [anthracyclines, trastuzumab, rituximab]), immuno-therapies (immune checkpoint inhibitors [ICI's]) or radiation (within 8 weeks of completion of radiation).29-31
* Ability to speak and understand English
* Capacity to walk at least 2 city blocks (~.2 miles) on a flat surface
* Expected survival beyond 6 months.
* Must have an assistant that will help perform the home-based testing activities

Exclusion Criteria:

If the patient meets any of these criteria they are excluded from the study:

* Uncontrolled hypertension (systolic blood pressure >190 mm Hg or diastolic blood pressure >100 mm Hg)
* Recent history of alcohol or drug abuse, inflammatory conditions such as lupus or inflammatory bowel disease, or another medical condition that might compromise safety or successful completion (unless approved by the participant's physician and the Principal Investigator) NOTE: In the setting of active inflammation, participation will not be approved. If chronic disease is present and stable as judged by the participant's physician and the PI, participation will be approved.
* Contraindications to MRI such as ferromagnetic cerebral aneurysm clips or other intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices (unless approved by the participant's physician and the Principal Investigator)
* Pregnant
* Unstable angina
* Contraindication for exercise training or testing
* Inability to exercise on a treadmill or stationary cycle
* Significant ventricular arrhythmias (>20 PVCs/min due to gating difficulty)
* Atrial fibrillation with uncontrolled ventricular response
* Acute myocardial infarction within 28 days
* Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Peak VO2 | At baseline and 6 months after study intervention
  An analysis of covariance (ANCOVA) model will be used to assess post-intervention group differences in VO2, adjusted for baseline peak VO2.

SECONDARY OUTCOMES:
Change in Peak Exercise Cardiac Output | At baseline and 6 months after study intervention
  Measured on a continuous scale and will be analyzed using a repeated measures ANCOVA (RMANCOVA) approach.
Change in Calculated A-V Oxygen Levels | At baseline and 6 months after study intervention
  Measured on a continuous scale and will be analyzed using a repeated measures ANCOVA (RMANCOVA) approach.
Changes in Measurements of Pre-exercise Left Ventricular Function | At baseline and 6 months after study intervention
  Measured on a continuous scale and will be analyzed using a repeated measures ANCOVA (RMANCOVA) approach.
Change in Neurocognitive Function - Hopkins Verbal Learning Test | At baseline and 6 months after study intervention
  The Hopkins Verbal Learning Test (HVLT-R) consists of memorization of a list of words to test the ability to recall immediately after memorization (immediate recall) and after a 20-minute delay (delayed recall). This test has three parts and two alternate forms. Total scores could range from 0 to 30. Lower raw scores indicate difficulties with the task.
Change in Neurocognitive Function - Controlled Oral Word Association Test (COWAT) | At baseline and 6 months after study intervention
  The Controlled Oral Word Association Test is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe (typically 60 seconds). COWAT is measured by calculating the total number of acceptable words produced for at the given letter of the alphabet. Errors and perseverations (word repetitions) are not included in this score.
Change in Neurocognitive Function - Digit Span-Backward Test | At baseline and 6 months after study intervention
  The digit span backward test is used to assess working memory. Participants are given a series of digits and asked to repeat them backward. The item score is the sum of the scores on the two trials for that item (range=0-2). The total raw score for backwards digit span is the sum of the item scores; maximum backwards digit span total raw score is 16 points.
Change in Neurocognitive Function - Trail Making Test | At baseline and 6 months after study intervention
  The Trail Making Test (TMT) asks patients to connect consecutive "targets" (numbers and/or letters) on a page arranged in a specific geometric pattern. Scoring is based on time taken to complete the test (e.g. 35 seconds yielding a score of 35) with lower scores being better.
Change in 6-Minute Walk Distance | At baseline, 3 months and 6 months after study intervention
  Measured on a continuous scale and will be analyzed using a repeated measures ANCOVA (RMANCOVA) approach.
Health-Related Quality of Life Questionnaire (FACT-Lym or FACT-B) | At baseline, 3 months and 6 months after study intervention
  FACT-Lym is 42-item questionnaire to assess the quality of life for lymphoma patients. 5-point Likert scale - 0 (not at all) to 4 (very much). Subscale domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Lymphoma Subscale. Some items are reverse scored. Subscales scores are added to get the total score. The higher the score, the better the quality of life. Scores can range from 0-168.
  FACT-B is a 37-item Functional Assessment of Cancer Therapy-Breast (FACT-B) that measures five domains of health-related quality of life in breast cancer patients. These include physical, social, emotional and functional well being on a Likert scale 0-4 with (not at all) to 4 (very much). The higher the score, the better quality of life. Scores can range from 0-148.
Fatigue Questionnaire | At baseline, 3 months and 6 months after study intervention
  Questionnaire to assess the difference in the level of fatigue participants experience will performing study interventions. 5-point Likert scale - 0 (not at all) to 4 (very much). The higher the score the higher level of fatigue participants experience. Score range 0-52.
Change in Physical Activity Levels - Godin Leisure Time Exercise Questionnaire | At baseline, 3 months and 6 months after study intervention
  The questionnaire is a 4-item measure used to classify participants' activity levels during a typical 7-day period based on how many times on average participants exercise more than 15 minutes during their free time of strenuous, moderate or mild exercise.
Change in Physical Function - Balance Test | At baseline, 3 months and 6 months after study intervention
  Participants will be asked to maintain balance for up to 30 seconds in three positions characterized by a progressive narrowing of the base support: heel of one foot beside the big toe of the other foot (semi-tandem position), heel of one foot in front of and touching the toes of the other foot (tandem position), and single leg stand.
Change in Physical Function - Chair Stand Test | At baseline, 3 months and 6 months after study intervention
  The repeated chair stand test will be performed using a straight-backed chair placed with its back against a wall. Participants will be first asked to stand from a sitting position without using their arms. If they can perform the task, they will then be asked to stand up and sit down five times as quickly as possible. The time to complete the task will be recorded.
Change in Physical Function - 4-Meter Walk Gait Speed Test | At baseline, 3 months and 6 months after study intervention
  The gait speed test will assess the participant's ability to walk 4 meters. Participants will be instructed to start at a marked walking course with toes touching the start line and when cued to start, will begin walking at their usual speed. The time to walk from the starting line to the end of the 4-meter walk will be recorded
Change in Physical Function - Grip Strength | At baseline, 3 months and 6 months after study intervention
  Grip strength will be assessed using an isometric handgrip dynamometer while the participant is seated with the head facing straight ahead. The elbow should be bent at a 90 degree angle and the wrist should be at the mid-prone position. The participant should exert maximally and quickly (about 1 second) and two trials should be made alternately with each hand, with at least 30 seconds between trials for the same hand (recorded in kilograms).

CONTACTS AND LOCATIONS:
Overall Officials: William Hundley, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No